CLINICAL TRIAL: NCT03428919
Title: The Effectiveness of Intracytoplasmic Sperm Injection Versus Conventional in Vitro Fertilization in Couples With Non-male Factor Infertility: a Randomized Controlled Trial
Brief Title: ICSI Versus Conventional IVF in Non-male Factor Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: An Sinh Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS/MD/17/12; CS/AS/17/10 (Other: An Sinh Hospital)
Record Dates: First submitted 2018-02-02; First posted 2018-02-12 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Infertility
Keywords: ICSI; Conventional IVF; Non-male factor
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracytoplasmic Sperm Injection (ICSI) (Active Comparator): All patients will be treated with a GnRH antagonist protocol. hCG (Ovitrelle 250 mg) will be used in the presence of at least three leading follicles of 17 mm. In women with ≥15 follicles ≥12 mm, 0,2 mg Triptorelin (Diphereline) will be used when there is at least two leading follicles of 17 mm. Oocyte retrieval will be performed 36 hours after triggering.
  Insemination will be performed by using ICSI, 3 - 4 hours after oocyte retrieval. OCCs will be stripped by using hyaluronidase. Only matured oocytes will be inseminated.
  Fertilization check will be performed at period of 16-18 hours after insemination. Embryo transfer will be performed on day 3 under ultrasound guidance. A maximum of 2 embryos will be transferred into the uterus. The remaining grade 1 and 2 embryos will be frozen.
  Interventions: Procedure: ICSI
- In Vitro Fertilization (IVF) (Active Comparator): All patients will be treated with a GnRH antagonist protocol. hCG (Ovitrelle 250 mg) will be used in the presence of at least three leading follicles of 17 mm. In women with ≥15 follicles ≥12 mm, 0,2 mg Triptorelin (Diphereline) will be used when there is at least two leading follicles of 17 mm. Oocyte retrieval will be performed 36 hours after triggering.
  Insemination will be performed by conventional IVF. Two hours after retrieval, collected OCCs will be inseminated for another 2 hours (100,000 motile sperm/ml). Inseminated OCCs will be cultured overnight in culture medium.
  Fertilization check will be performed at period of 16-18 hours after insemination. Embryo transfer will be performed on day 3. A maximum of 2 embryos will be transferred. The remaining grade 1-2 embryos will be frozen.
  Interventions: Procedure: IVF

INTERVENTIONS:
Procedure: ICSI — In ICSI group, insemination will be performed by using ICSI, 3 - 4 hours after oocyte retrieval. OCCs will be stripped by using hyaluronidase. Only matured oocytes will be inseminated.
  Arms: Intracytoplasmic Sperm Injection (ICSI)
Procedure: IVF — In IVF group, insemination will be performed by conventional IVF. Two hours after retrieval, collected OCCs will be inseminated for another 2 hours, at a concentration of 100,000 motile sperm/ml. Inseminated OCCs will be cultured overnight in culture medium.
  Arms: In Vitro Fertilization (IVF)

SUMMARY:
Conventionally, ICSI was initially developed and has been shown to be an effective treatment for male factor infertility. It is increasingly being used for patients without a male factor diagnosis, despite the lack of clinical evidence to support its use. Moreover, ICSI is an invasive and expensive procedure. This multi-center, randomized, controlled, parallel-group trial will be conducted to compare the effectiveness of ICSI versus conventional IVF in infertile couples scheduled for IVF treatment, in whom the male partner has normal sperm.

DETAILED DESCRIPTION:
All patients undergoing IVF/ICSI will be treated with a GnRH antagonist protocol. Recombinant FSH (Puregon, MSD) will be given on day 2 or day 3 of menstrual cycle for 5 days. The starting dose is individualized for each patient based on the following criteria: AMH <0.7 ng/mL, dose 300 IU/day; AMH 0.7-2.1 ng/mL, dose 200 IU/day; AMH >2.1 ng/mL, dose 150 IU/day. After that, investigators can titrate the dose based on their clinical judgment. Follicular development will be monitored by ultrasound scanning and measurement of estradiol and progesterone levels, starting on day 5 of stimulation. Scanning and hormonal measurement will be repeated every 2 to 3 days, depending on the size of follicles. An antagonist is routinely used on day 5 until the day of triggering. Criteria for triggering, by hCG (Ovitrelle 250 mg, Merck, Germany) will be the presence of at least three leading follicles of 17 mm. In women with excessive follicular response (≥15 follicles ≥12 mm), 0,2 mg Triptorelin (Diphereline, Ipsen Beaufour, France) will be used when there are at least two leading follicles of 17 mm. Oocyte retrieval will be performed 36 hours after triggering.

Randomization and allocation of participants to study groups will be performed on the day of egg pick up, after having obtained the semen from the husband. Eligible participants that have provided informed consent will be randomised to either ICSI or conventional IVF.

In ICSI group, insemination will be performed by using ICSI, 3 - 4 hours after oocyte retrieval. OCCs will be stripped by using hyaluronidase. Only matured oocytes will be inseminated.

In conventional IVF group, insemination will be performed by conventional IVF. Two hours after retrieval, collected OCCs will be inseminated for another 2 hours, at a concentration of 100,000 motile sperm/ml. Inseminated OCCs will be cultured overnight in culture medium.

In both groups, fertilization check will be performed under inverted microscope at period of 16-18 hours after insemination. On day 3, embryo evaluation will be performed at fixed time point 66±2 hours after fertilization, using the Istanbul consensus. Embryo transfer will be performed on day 3 under ultrasound guidance. A maximum of 2 embryos will be transferred into the uterus. The remaining grade 1 and 2 embryos will be frozen. Luteal-phase support will be done with estradiol (Valiera 2mg) 8mg/day and vaginal progesterone 800mg/day (Cyclogest 400mg) until 7th week of gestation.

If there are contra-indications for fresh embryo transfer, a freeze-all strategy will be applied, using Cryotech technique. Indications for freeze-all include: risk of ovarian hyperstimulation syndrome (OHSS), premature progesterone rise (≥1.5 ng/ml), thin endometrium (<7 mm), fluid in cavity on day of embryo transfer, endometrial polyp, hydrosalpinx that have not removed before oocyte retrieval.

In the next cycle, endometrium will be prepared by using estradiol (Valiera 2 mg, 8 mg/day) orally, starting from day 2-3 of menstrual cycle. When the endometrium thickness reaches 8 mm or more, patients will start using progesterone vaginally (Cyclogest 400 mg, 800 mg/day). Embryo transfer will be performed 3 days after using progesterone. On the day of embryo transfer, embryos will be thawed. In the frozen/thawed cycle, the best embryos will be utilized first, as in fresh transfer. Two hours after thawing, a maximum of 2 surviving embryos will be transferred into the uterus under ultrasound guidance. Luteal phase support will be provided with estradiol (Valiera 2mg) 8mg/day and vaginal progesterone 800 mg/day (Cyclogest 400 mg) until the seventh week of gestation.

In both groups, clinicians who perform embryo transfer, either fresh or frozen cycles, will be blinded to the intervention.

A serum hCG will be measured 2 weeks after embryo transferred, and if positive, an ultrasound scan of the uterus will be performed at gestational weeks 7 and 12. At 11 - 12 weeks of gestation, participants will be referred to the Outpatient clininc, O&G Department, My Duc hospital or An Sinh hospital for prenatal care until giving birth.

ELIGIBILITY:
Inclusion Criteria:

* Having ≤ 2 IVF/ICSI cycles
* Total sperm count and motility are normal (WHO, 2010)
* Antagonist protocol
* Agree to have ≤ 2 embryos transferred
* Not participating in another IVF study at the same time

Exclusion Criteria:

* In-vitro maturation (IVM) cycles
* Using frozen semen
* Poor fertilization in previous cycle (≤ 25%)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1064 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy resulting in live birth after the first embryo transfer of the started treatment cycle. | At 12 weeks of gestation
  Live birth is defined as the birth of at least one newborn after 24 weeks' gestation that exhibits any sign of life (twin will be a single count).
  For the timing of this occur, ongoing pregnancy will be used, conditional on the fact that this ongoing pregnancy results in live birth.

SECONDARY OUTCOMES:
Fertilization rate per oocyte inseminated/injected | At 16-18 hours after injected or 17-19 hours after inseminated
  Fertilization is defined as the appearance of 2 PN
Fertilization rate per oocyte retrieved | At 16-18 hours after injected or 17-19 hours after inseminated
  Fertilization is defined as the appearance of 2 PN
Abnormal fertilization rate | At 16-18 hours after injected or 17-19 hours after inseminated
  Abnormal fertilization is defined as the appearance of 1PN or ≥3 PN
Total fertilization failure rate | At 16-18 hours after injected or 17-19 hours after inseminated
  Total fertilization is defined as the absence of any zygotes with 2PN
Number of embryos on day 3 | 3 days after oocytes pick-up day in IVF/ICSI
  Number of embryos on day 3
Number of good quality embryo on day 3 | 3 days after oocytes pick-up day in IVF/ICSI
  Numbers of embryos on day 3 with good quality
Number of embryo freezing on day 3 | 3 days after oocytes pick-up day in IVF/ICSI
  Number of embryos freezing on day 3
Positive pregnancy test | 14 days after embryo transfer
  Positive pregnancy test is defined as a serum human chorionic gonadotropin level greater than 25 mIU/mL after the completion of the first transfer
Clinical pregnancy | At 7 weeks' gestation
  Clinical pregnancy is defined as the presence of at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity, after the completion of the first transfer
Implantation rate | At 3 weeks after embryo transferred
  Implantation rate is defined as the number of gestational sacs per number of embryos transferred after the completion of the first transfer
Ongoing pregnancy | At 12 weeks' gestation
  Ongoing pregnancy is defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond, after the completion of the first transfer
Cumulative ongoing pregnancy | At 12 weeks' gestation at 12 months after randomization. After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative ongoing pregnancy rate.
  Ongoing pregnancy is defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond, after transfer of all embryos from the started treatment cycle.
Ongoing pregnancy resulting in live birth obtained from all embryos from the first started treatment cycle | 12 weeks of gestation at 12 months after randomization
  Live birth is defined as the birth of at least one newborn after 24 weeks' gestation that exhibits any sign of life (twin will be a single count).
Time from randomization to ongoing pregnancy | 12 weeks of gestation after the completion of first transfer
  Time from randomization to ongoing pregnancy after the completion of the first transfer
Ovarian hyperstimulation syndrome (OHSS) | At 10 days after hCG injection and 14 days after embryo transfer
  Symptoms of OHSS
Ectopic pregnancy | At 12 weeks of gestation after the completion of the first transfer
  A pregnancy in which implantation takes place outside the uterine cavity after completion of the first transfer
Ectopic pregnancy | At 12 weeks of gestation at 12 months after randomization.
  A pregnancy in which implantation takes place outside the uterine cavity after transfer of all embryos from the started treatment cycle.
Miscarriage | At 24 weeks of gestation after the completion of the first transfer
  The loss of a clinical pregnancy at 24 weeks of gestation after the completion of the first transfer
Miscarriage | At 24 weeks of gestation at 12 months after the randomization.
  The loss of a clinical pregnancy at 24 weeks of gestation after the completion transfer of all embryos from the started treatment cycle
Multiple pregnancy | 7 weeks' gestation after the completion of the first transfer
  Multiple pregnancy is explained as two or more gestational sacs or positive heart beats by transvaginal sonography, after the completion of the first transfer
Multiple pregnancy | 7 weeks' gestation at 12 months after randomization
  Multiple pregnancy is explained as two or more gestational sacs or positive heart beats by transvaginal sonography, after the completion transfer of all embryos from the started treatment cycle
Multiple delivery | At birth, after the completion of the first transfer
  Multiple delivery is defined as birth of more than one baby beyond 24 weeks, after the completion of the first transfer
Multiple delivery | At birth at 12 months after randomization
  Multiple delivery is defined as birth of more than one baby beyond 24 weeks, after the completion transfer of all embryos from the started treatment cycle
Gestational diabetes mellitus | At 24 weeks of gestation after the completion of the first transfer
  Development of diabetes during pregnancy
Gestational diabetes mellitus | At 24 weeks of gestation at 12 months after randomization
  Development of diabetes during pregnancy
Hypertensive disorders of pregnancy | From 20 weeks of gestation up to at birth after the completion of the first transfer
  Hypertensive disorders of pregnancy will include pregnancy induced hypertension (PIH); pre-eclampsia (PET) and eclampsia)
Hypertensive disorders of pregnancy | From 20 weeks of gestation up to at birth at 12 months after randomization
  Hypertensive disorders of pregnancy will include pregnancy induced hypertension (PIH); pre-eclampsia (PET) and eclampsia)
Antepartum haemorrhage | From 20 weeks of gestation up to at birth, after the completion of the first transfer
  Including placenta previa, placenta accreta and unexplained
Antepartum haemorrhage | From 20 weeks of gestation up to at birth, at 12 months after randomization
  Including placenta previa, placenta accreta and unexplained
Gestational age at delivery | At birth, after the completion of the first transfer
  Gestational age at delivery
Gestational age at delivery | At birth, at 12 months after randomization
  Gestational age at delivery
Preterm delivery | At birth, after the completion of the first transfer
  Preterm delivery is defined as any delivery at <24, <28, <32, <37 completed weeks' gestation
Preterm delivery | At birth, at 12 months after randomization
  Preterm delivery is defined as any delivery at <24, <28, <32, <37 completed weeks' gestation
Spontaneous preterm birth | At birth, after the completion of the first transfer
  Spontaneous preterm birth is defined as delivery spontaneously at <24, <28, <32, <37 completed weeks
Spontaneous preterm birth | At birth, at 12 months after randomization
  Spontaneous preterm birth is defined as delivery spontaneously at <24, <28, <32, <37 completed weeks
Iatrogenic preterm birth | At birth, after the completion of the first transfer
  Iatrogenic preterm birth is defined as delivery non-spontaneously at <24, <28, <32, <37 completed weeks
Iatrogenic preterm birth | At birth, at 12 months after randomization
  Iatrogenic preterm birth is defined as delivery non-spontaneously at <24, <28, <32, <37 completed weeks
Birth weight | At birth, after the completion of the first transfer
  Weight of newborn
Birth weight | At birth, at 12 months after randomization
  Weight of newborn
Low birth weight | At birth, after the completion of the first transfer
  Low birth weight is defined as <2500 gm
Low birth weight | At birth, at 12 months after randomization
  Low birth weight is defined as <2500 gm
Very low birth weight | At birth, after the completion of the first transfer
  Very low birth weight is defined as <1500 gm
Very low birth weight | At birth, at 12 months after randomization
  Very low birth weight is defined as <1500 gm
High birth weight | At birth, after the completion of the first transfer
  High birth weight is defined as >4000 gm
High birth weight | At birth, at 12 months after randomization
  High birth weight is defined as >4000 gm
Very high birth weight | At birth, after the completion of the first transfer
  Very high birth weight is defined as >4500 gm
Very high birth weight | At birth, at 12 months after randomization
  Very high birth weight is defined as >4500 gm
Large for gestational age | At birth, after the completion of the first transfer
  Large for gestational age is defined as birth weight >90th percentile
Large for gestational age | At birth, at 12 months after randomization
  Large for gestational age is defined as birth weight >90th percentile
Small for gestational age | At birth, after the completion of the first transfer
  Small for gestational age is defined as birth weight <10th percentile
Small for gestational age | At birth, at 12 months after randomization
  Small for gestational age is defined as birth weight <10th percentile
Congenital anomaly diagnosed at birth | At birth, after the completion of the first transfer
  Any congenital anomaly will be included
Congenital anomaly diagnosed at birth | At birth, at 12 months after randomization
  Any congenital anomaly will be included
Admission to NICU | 7 days after delivery after the completion of the first transfer
  The admittance of the newborn to NICU
Admission to NICU | 7 days after delivery, at 12 months after randomization
  The admittance of the newborn to NICU
Genetic and epigenetic analysis of newborn | 1 day (Prior to the initiation of IVF/IVM) and 1 day ( at the time of delivery)
  Maternal whole blood; newborn's materials including cord blood, neonatal buccal smear, and placental tissue will be collected. Data will be collected for a supplementary analysis and will be reported in a separated paper.
Cost-effectiveness | Two year after randomization
  Including direct and indirect costs; costs related to complications treatment. Cost data will be collected for a supplementary analysis and will be reported in a separated paper.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Dang Q Vinh, Hochiminh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pham TD, Dang VQ, Ho VNA, Tran CT, Nguyen DTP, Vuong LN, Ho TM, Mol BW, Wang R. Intracytoplasmic sperm injection versus conventional in vitro fertilization in infertile couples with normal total sperm count and motility: does sperm morphology matter? Hum Reprod. 2025 Jan 1;40(1):23-29. doi: 10.1093/humrep/deae252. PMID 39547931
- [Derived] Nguyen NA, Nguyen NT, Tran VTT, Vo TTM, Uong TS, Nguyen HT, Nguyen NT, Nguyen DL, Pham TD, Nguyen DTN, Ho TM, Vuong LN. Developmental outcomes of children born through ICSI versus conventional IVF (cIVF) in couples with non-male factor infertility. Hum Reprod. 2024 Jun 5:deae120. doi: 10.1093/humrep/deae120. Online ahead of print. PMID 38840410
- [Derived] Dang VQ, Vuong LN, Luu TM, Pham TD, Ho TM, Ha AN, Truong BT, Phan AK, Nguyen DP, Pham TN, Pham QT, Wang R, Norman RJ, Mol BW. Intracytoplasmic sperm injection versus conventional in-vitro fertilisation in couples with infertility in whom the male partner has normal total sperm count and motility: an open-label, randomised controlled trial. Lancet. 2021 Apr 24;397(10284):1554-1563. doi: 10.1016/S0140-6736(21)00535-3. PMID 33894833
- [Derived] Dang VQ, Vuong LN, Ho TM, Ha AN, Nguyen QN, Truong BT, Pham QT, Wang R, Norman RJ, Mol BW. The effectiveness of ICSI versus conventional IVF in couples with non-male factor infertility: study protocol for a randomised controlled trial. Hum Reprod Open. 2019 Mar 27;2019(2):hoz006. doi: 10.1093/hropen/hoz006. eCollection 2019. PMID 30937394